CLINICAL TRIAL: NCT05459766
Title: Effects of a Perioperative Action Observation and Motor Imagery Training in Patients Undergoing Total Knee Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLF22/06
Record Dates: First submitted 2022-07-12; First posted 2022-07-15 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Total Knee Arthoplasty

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AO+MI (Experimental): Video-clips observation representing motor contents, followed by motor imagery (12 minutes a day per 3 days).
  Interventions: Behavioral: Action observation and motor imagery
- CTRL (Active Comparator): Usual care, consisting of preoperative education.
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: Action observation and motor imagery — Observation and imagination of functional tasks that will be performed during the postoperative rehabilitation program.
  Arms: AO+MI
Behavioral: Usual care — Participants will be educated about the postoperative rehabilitation program
  Arms: CTRL

SUMMARY:
The study is aimed at investigating the effects of action observation and motor imagery training in patients undergoing total knee arthroplasty. Fifty participants will be enrolled during hospital admission and randomized into 2 groups (AO+MI and CTRL groups). AO+MI will undergo 12-minute AO+MI intervention for 3 days (preoperative day, first and second postoperartive days), whereas CTRL group will undergo usual care. At baseline, first and third postoperative days, participants will be assessed for mobility, pain, range of motion, quadriceps acrivation failure and patient's bady-pain representation by a blinded operator.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for total knee arthroplasty
* age greater or equal to 18 years old
* ability to walk independently.

Exclusion Criteria:

* previous total knee arthoplasty on the contralateral side
* revision surgery
* dementia
* musculoskeletal and neurological disorders influencing functional recovery
* visual or auditory deficits.
* postoperative complications
* weight bearing restrictions
* lack of walking independency within the second postoperative day.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2023-01-31 (Estimated); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
Changes in functional mobility | At baseline, at 1 day and 3 days after surgery
  It will be assessed using the Timed Up and Go test

SECONDARY OUTCOMES:
Changes in active and passive knee range of motion | At baseline, at 1 day and 3 days after surgery
  It will be assessed using an inertial measurement unit
Changes in perceived pain | At baseline and 3 days after surgery
  It will be assessed using Numerical Rating Scale (0-10 points), where 0 means no pain and 10 means maximum pain.
Changes in body pain representation at the level of the knee joint | At baseline and 3 days after surgery
  It will be assessed using the Pain Drawing Body Chart
Changes in quadriceps activation failure | At baseline, at 1 day and 3 days after surgery
  It will be assessed using the Quadricpes Activation Battery

IPD SHARING:
Plan to Share IPD: No